CLINICAL TRIAL: NCT01755767
Title: A Phase 3, Randomized, Double-Blind Study of Tivantinib (ARQ 197) in Subjects With MET Diagnostic-High Inoperable Hepatocellular Carcinoma Treated With One Prior Systemic Therapy
Brief Title: Study of Tivantinib in Subjects With Inoperable Hepatocellular Carcinoma (HCC) Who Have Been Treated With One Prior Therapy
Acronym: METIV-HCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARQ197-A-U303; 2012-003308-10 (EudraCT Number)
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Results first posted 2020-07-15 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: MET diagnostic-high; Unresectable; Hepatocellular; Carcinoma; c-Met inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma | interventions — ARQ 197

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tivantinib 240 mg BID Cohort (Experimental): The tivantinib dosage of 240 mg tablets administered by mouth twice daily (BID), once in the morning and once in the evening, with food, for a total daily dose of 480 mg.
  Interventions: Drug: Tivantinib
- Tivantinib 120 mg BID Cohort (Experimental): Tivantinib 120 mg is administered by oral tablet BID, once in the morning and once in the evening, with food, for a total daily dose of 240 mg (amended dosing group; primary analysis group).
  Interventions: Drug: Tivantinib
- Placebo Matching 240 mg BID Cohort (Placebo Comparator): Matching placebo is administered by oral tablet(s) BID, once in the morning and once in the evening, with food.
  Interventions: Drug: Placebo
- Placebo Matching 120 mg BID Cohort (Placebo Comparator): Matching placebo is administered by oral tablet(s) BID, once in the morning and once in the evening, with food.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tivantinib — Tivantinib tablets
  Other Names: ARQ197
  Arms: Tivantinib 120 mg BID Cohort; Tivantinib 240 mg BID Cohort
Drug: Placebo — Matching placebo tablets
  Other Names: Placebo comparator
  Arms: Placebo Matching 120 mg BID Cohort; Placebo Matching 240 mg BID Cohort

SUMMARY:
The purpose of this study is to determine if tivantinib (ARQ 197) is effective in treating patients with MET diagnostic-high hepatocellular carcinoma (liver cancer) who have already been treated once with another therapy.

DETAILED DESCRIPTION:
Expression of c-Met in tumors correlates with aggressive hepatocellular carcinoma (HCC) features. Overexpression of the receptor in tumor samples or high level of blood HGF in subjects is related to higher recurrence rate after surgery for HCC, while high c-Met expression correlates with shorter survival in HCC subjects. In summary, c-Met holds an important prognostic role in the natural history of HCC. This Phase 3 study in MET Diagnostic-High inoperable HCC subjects has been designed based on the results from the randomized, controlled Phase 2 study conducted by ArQule, Inc. with tivantinib versus placebo in subjects with MET Diagnostic-High inoperable HCC who have failed one prior systemic therapy, mentioned above. The purpose of this study is to confirm the efficacy of tivantinib in MET Diagnostic-High HCC subjects who were previously treated with one systemic therapy, and to further evaluate the safety profile of the experimental drug in this subject population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HCC that is inoperable (where surgery is not indicated due to disease extension, co-morbidities, or other technical reasons), and not eligible for local therapy
* MET Diagnostic-High tissue reported by the central authorized laboratory using archival or recent biopsy tumor samples
* Received at least 4 weeks of one prior sorafenib containing systemic therapy and then experienced documented radiographic disease progression; or inability to tolerate prior therapy received for at least a minimum period of time.
* Discontinued prior systemic treatment or any investigational drug for at least 2 weeks (14 days) or for at least 3 weeks for IV anti-cancer drugs, prior to the study randomization
* Local or loco-regional therapy (i.e., surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation) must have been completed >= 4 weeks prior to randomization
* Measurable disease as defined by the RECIST v1.1.

Exclusion Criteria:

* More than 1 prior systemic regimen (prior MET inhibitors/antibodies are not allowed; experimental systemic therapy for inoperable HCC given before or after sorafenib counts as separate regimen and is not allowed)
* Child-Pugh B-C cirrhotic status based on clinical findings and laboratory results
* Previous or concurrent cancer that is distinct from HCC in primary site or histology, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, and superficial bladder tumors. Any cancer curatively treated more than 3 years prior to enrollment is permitted.
* History of congestive heart failure defined as Class II to IV per New York Heart Association (NYHA) classification within 6 months prior to study entry; active coronary artery disease (CAD); clinically significant bradycardia or other uncontrolled, cardiac arrhythmia defined as greater than or equal to Grade 3 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), or uncontrolled hypertension; myocardial infarction occurring within 6 months prior to study entry (myocardial infarction occurring more than 6 months prior to study entry is permitted)
* Active clinically serious infections defined as >= Grade 3 according to NCI CTCAE
* Any medical, psychological, or social conditions, particularly if unstable, including substance abuse, that may, in the opinion of the Investigator, interfere with the subject's safety or participation in the study, protocol compliance, or evaluation of the study results
* Known human immunodeficiency virus (HIV) infection
* Blood or albumin transfusion within 5 days prior to the blood draw being used to confirm eligibility
* Concomitant interferon therapy or therapies for active Hepatitis C virus (HCV) infection
* Pregnancy or breast-feeding
* History of liver transplant
* Inability to swallow oral medications
* Clinically significant gastrointestinal bleeding occurring <= 4 weeks prior to randomization
* Pleural effusion or clinically evident (visible or palpable) ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2012-12-27 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (112):
- United States (20):
  - Tucson, Arizona
  - Los Angeles, California
  - Orange, California
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Chicago, Illinois
  - Westwood, Kansas
  - New Orleans, Louisiana
  - Scarborough, Maine
  - Boston, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Hackensack, New Jersey
  - New York, New York
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Galveston, Texas
  - Houston, Texas
  - Seattle, Washington
- Argentina (3):
  - Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Buenos Aires, Buenos Aires F.D.
  - Pilar
- Australia (4):
  - Camperdown, New South Wales
  - Heidelberg, Victoria
  - Melbourne, Victoria
  - Nedlands, Western Australia
- Austria (4):
  - Graz
  - Innsbruck
  - Linz
  - Vienna
- Belgium (4):
  - Brussels
  - Ghent
  - Leuven
  - Liège
- Brazil (4):
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
  - Barretos
  - Rio de Janeiro
- Canada (2):
  - Vancouver, British Columbia
  - Toronto, Ontario
- France (14):
  - Amiens
  - Bordeaux
  - Caen
  - Clichy
  - Créteil
  - Grenoble
  - Lille
  - Marseille
  - Montpellier
  - Paris
  - Reims
  - Rennes
  - Toulouse
  - Villejuif
- Germany (18):
  - Aachen
  - Berlin
  - Bonn
  - Düsseldorf
  - Essen
  - Frankfurt am Main
  - Hamburg
  - Hanover
  - Heidelberg
  - Leipzig
  - Magdeburg
  - Mainz
  - Munich
  - München
  - Regensburg
  - Tübingen
  - Ulm
  - Würzburg
- Italy (18):
  - Meldola, Forli-Cesena
  - Rozzano, Milano
  - Orbassano (TO), Torino
  - Benevento
  - Bergamo
  - Bologna
  - Catania
  - Florence
  - Milan
  - Modena
  - Napoli
  - Padua
  - Parma
  - Pavia
  - Pisa
  - Reggio Emilia
  - Roma
  - Turin
- Amsterdam, Netherlands
- Auckland, New Zealand
- Portugal (3):
  - Lisbon
  - Porto
  - Vila Real
- Spain (12):
  - Santiago de Compostela, A Coruña
  - Majadahonda, Madrid
  - Pamplona, Navarre
  - Oviedo, Principality of Asturias
  - Alicante
  - Barcelona
  - Córdoba
  - Madrid
  - Sabadell
  - Santander
  - Valencia
  - Zaragoza
- Sweden (2):
  - Gothenburg
  - Stockholm
- Switzerland (2):
  - Bern
  - Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rimassa L, Assenat E, Peck-Radosavljevic M, Pracht M, Zagonel V, Mathurin P, Rota Caremoli E, Porta C, Daniele B, Bolondi L, Mazzaferro V, Harris W, Damjanov N, Pastorelli D, Reig M, Knox J, Negri F, Trojan J, Lopez Lopez C, Personeni N, Decaens T, Dupuy M, Sieghart W, Abbadessa G, Schwartz B, Lamar M, Goldberg T, Shuster D, Santoro A, Bruix J. Tivantinib for second-line treatment of MET-high, advanced hepatocellular carcinoma (METIV-HCC): a final analysis of a phase 3, randomised, placebo-controlled study. Lancet Oncol. 2018 May;19(5):682-693. doi: 10.1016/S1470-2045(18)30146-3. Epub 2018 Apr 3. PMID 29625879

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 383 participants who met all inclusion criteria and no exclusion criteria were randomized to treatment. One participant in the tivantinib 120 mg BID cohort was randomized but did not receive treatment.
Pre-assignment Details: Eligible participants were randomly assigned on a 2:1 basis to either tivantinib or placebo. Initially, the tivantinib dosage of 240 mg was selected on the basis of efficacy and tolerability established in Phase 1 and Phase 2 studies.
Groups:
- Tivantinib 240 mg BID Cohort: Participants who received tivantinib 240 mg tablets administered by mouth twice daily (BID), once in the morning and once in the evening, with food, for a total daily dose of 480 mg.
- Placebo Matching 240 mg BID Cohort; Placebo Matching 120 mg BID Cohort: Participants who received matching placebo tablets administered by mouth twice daily (BID), once in the morning and once in the evening, with food.
- Tivantinib 120 mg BID Cohort: Participants who received tivantinib 120 mg tablets administered by mouth twice daily (BID), once in the morning and once in the evening, with food, for a total daily dose of 240 mg (amended dosing group; primary analysis group).
Period: Overall Study
Arm/Group | Tivantinib 240 mg BID Cohort | Placebo Matching 240 mg BID Cohort | Tivantinib 120 mg BID Cohort | Placebo Matching 120 mg BID Cohort
Started | 28 | 15 | 226 | 114
Completed | 0 | 0 | 0 | 0
Not Completed | 28 | 15 | 226 | 114
Not completed — Progressive Disease | 8 | 7 | 91 | 43
Not completed — Clinical Disease Progression | 4 | 2 | 29 | 20
Not completed — Radiographic Disease Progression | 9 | 4 | 44 | 27
Not completed — Adverse Event | 6 | 0 | 28 | 11
Not completed — Death | 1 | 2 | 15 | 4
Not completed — Subject Decision | 0 | 0 | 10 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Other | 0 | 0 | 2 | 3
Not completed — Ongoing Treatment as of 06 Jan 2017 | 0 | 0 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics are reported in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tivantinib 240 mg BID Cohort | Placebo Matching 240 mg BID Cohort | Tivantinib 120 mg BID Cohort | Placebo Matching 120 mg BID Cohort | Total
Number analyzed (Participants) | 28 | 15 | 225 | 114 | 382
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 5 | 98 | 50 | 164
  >=65 years | 17 | 10 | 127 | 64 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (9.3) | 64.9 (7.4) | 65.6 (10.2) | 64.7 (10.2) | 64.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 27 | 7 | 38
  Male | 24 | 15 | 198 | 107 | 344
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 2
  Asian | 1 | 0 | 8 | 7 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 11 | 1 | 12
  White | 27 | 15 | 161 | 86 | 289
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 43 | 20 | 63

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival (OS) Following Treatment With Tivantinib 120 mg BID Compared to Placebo Group in Participants With MET Diagnostic-High Inoperable Hepatocellular Carcinoma (HCC) Treated With One Prior Systemic Therapy
Description: Overall survival (OS) is defined as the time from randomization to the date of death. The rate of OS (percentage of participants still alive) was determined only in the tivantinib 120 mg BID cohort.
Time Frame: within 36 months
Population: Overall survival was assessed in the Intent-to-Treat Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tivantinib 120 mg BID Cohort | Placebo Matching 120 mg BID Cohort
Number analyzed (Participants) | 226 | 114
months | 8.4 [6.8 to 10.0] | 9.1 [7.3 to 10.4]
Statistical Analysis 1: Comparison: Tivantinib 120 mg BID Cohort; Test type: Superiority; p = 0.8006, Log Rank; Stratified log rank between treatment arms adjusted for stratification factors: vascular invasion, extra-hepatic spread, and alpha fetoprotein level
Statistical Analysis 2: Comparison: Tivantinib 120 mg BID Cohort vs Placebo Matching 120 mg BID Cohort; Test type: Superiority; p = 0.8061, Regression, Cox; Stratified Cox Regression between treatment arms adjusted for factors: vascular invasion, extra-hepatic spread, and alpha fetoprotein level; Hazard Ratio (HR) = 0.9682, 95% CI 2-sided [0.7483 to 1.2529]

2. Primary Outcome: Overall Survival (OS) Rate At Different Time Points Following Treatment With Tivantinib 120 mg BID Compared to Placebo Group in Participants With MET Diagnostic-High Inoperable Hepatocellular Carcinoma (HCC) Treated With One Prior Systemic Therapy
Description: as for outcome 1
Time Frame: within 36 months
Population: Overall survival was assessed in the Intent-to-Treat Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants still alive
Arm/Group | Tivantinib 120 mg BID Cohort | Placebo Matching 120 mg BID Cohort
Number analyzed (Participants) | 226 | 114
percentage of participants still alive
  Overall survival at 3 months | 86.6 [81.4 to 90.5] | 85.9 [78.0 to 91.1]
  Overall survival at 6 months | 61.2 [54.5 to 67.2] | 70.8 [61.5 to 78.3]
  Overall survival at 9 months | 46.9 [40.2 to 53.3] | 50.5 [40.9 to 59.2]
  Overall survival at 12 months | 36.6 [30.3 to 42.9] | 38.0 [29.1 to 46.9]
  Overall survival at 18 months | 25.1 [19.4 to 31.2] | 21.9 [14.3 to 30.5]
  Overall survival at 24 months | 16.2 [11.0 to 22.3] | 12.2 [5.9 to 20.8]

3. Secondary Outcome: Progression-free Survival Following Treatment With Tivantinib 120 mg BID Compared to Placebo Group in Participants With MET Diagnostic-High Inoperable Hepatocellular Carcinoma (HCC) Treated With One Prior Systemic Therapy (ITT Population)
Description: Progression-free survival (PFS) is defined as the time from the date of randomization to the date of the first radiographic disease progression or death due to any cause. The rate of PFS (percentage of participants still alive without disease progression) was determined only in the tivantinib 120 mg BID cohort.
Time Frame: within 10 months
Population: PFS was assessed in the Intent-to-Treat Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tivantinib 120 mg BID Cohort | Placebo Matching 120 mg BID Cohort
Number analyzed (Participants) | 226 | 114
months | 2.1 [1.9 to 3.0] | 2.0 [1.9 to 3.6]
Statistical Analysis 1: Comparison: Tivantinib 120 mg BID Cohort vs Placebo Matching 120 mg BID Cohort; Test type: Superiority; p = 0.7509, Log Rank; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Tivantinib 120 mg BID Cohort vs Placebo Matching 120 mg BID Cohort; Test type: Superiority; p = 0.7160, Regression, Cox; [statistical method as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.9557, 95% CI 2-sided [0.7487 to 1.2200]

4. Secondary Outcome: Treatment-Emergent Adverse Events Reported (>20% in Tivantinib Cohort) Following Treatment With Tivantinib Compared With Placebo in Participants With MET Diagnostic-High Inoperable Hepatocellular Carcinoma (HCC) Treated With One Prior Systemic Therapy
Description: Treatment-emergent adverse events (TEAEs) are reported for the tivantinib 120 mg BID cohort group.
Time Frame: Baseline to 30 days after last dose, up to approximately 4 years
Population: TEAEs were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Tivantinib 120 mg BID Cohort | Placebo Matching 120 mg BID Cohort
Number analyzed (Participants) | 225 | 114
Participants
  Any TEAEs | 214 | 108
  Gastrointestinal Disorders | 159 | 84
  General Disorders & Administration Site Conditions | 146 | 75
  Musculoskeletal and Connective Tissue Disorders | 75 | 34
  Respiratory, Thoracic, and Mediastinal Disorders | 70 | 32
  Metabolism and Nutrition Disorders | 65 | 30
  Blood and Lymphatic System Disorders | 64 | 27
  Nervous System Disorders | 60 | 27
  Infections and Infestations | 58 | 33
  Skin and Subcutaneous Tissue Disorders | 57 | 38
  Investigations | 55 | 36
  Cardiac Disorders | 52 | 13

5. Secondary Outcome: Treatment-Emergent Adverse Events Reported (>20% in Tivantinib Cohort) Following Treatment With Tivantinib Compared With Placebo in Participants With MET Diagnostic-High Inoperable Hepatocellular Carcinoma (HCC) Treated With One Prior Systemic Therapy
Description: Treatment-emergent adverse events (TEAEs) are reported for the tivantinib 240 mg BID cohort group.
Time Frame: Baseline to 30 days after last dose, up to approximately 4 years
Population: TEAEs were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Tivantinib 240 mg BID Cohort: Participants who received tivantinib 240 mg tablets administered by mouth twice daily (BID), once in the morning and once in the evening, with food, for a total daily dose of 480 mg (amended dosing group; primary analysis group).
Arm/Group | Tivantinib 240 mg BID Cohort | Placebo Matching 240 mg BID Cohort
Number analyzed (Participants) | 28 | 15
Participants
  Any TEAEs | 28 | 14
  Blood and Lymphatic System Disorders | 20 | 4
  Gastrointestinal Disorders | 20 | 12
  General Disorders & Administration Site Conditions | 19 | 9
  Investigations | 11 | 8
  Respiratory, Thoracic, and Mediastinal Disorders | 8 | 4
  Infections and Infestations | 7 | 3
  Skin and Subcutaneous Tissue Disorders | 7 | 3
  Cardiac Disorders | 7 | 0
  Metabolism and Nutrition Disorders | 6 | 5

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from baseline to 30 days after the last dose up to approximately 4 years.
Description: Treatment-emergent AEs (TEAEs) were defined as those AEs that occurred, having been absent before the study, or worsen in severity after the initiation of study treatment administration and started no later than 30 days after the end of treatment.
Arm/Group | Tivantinib 240 mg BID Cohort | Placebo Matching 240 mg BID Cohort | Tivantinib 120 mg BID Cohort | Placebo Matching 120 mg BID Cohort
All-Cause Mortality (participants affected / at risk) | 28/28 | 14/15 | 180/225 | 94/114
Serious Adverse Events (participants affected / at risk) | 17/28 | 10/15 | 103/225 | 51/114
Other Adverse Events (participants affected / at risk) | 17/28 | 10/15 | 214/225 | 108/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tivantinib 240 mg BID Cohort (N=28) | Placebo Matching 240 mg BID Cohort (N=15) | Tivantinib 120 mg BID Cohort (N=225) | Placebo Matching 120 mg BID Cohort (N=114)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 2 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 4
Ascites (Gastrointestinal disorders) | 0 | 2 | 7 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 8 | 2
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 2 | 6 | 3
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
Device malfunction (General disorders) | 0 | 0 | 0 | 1
Disease progression (General disorders) | 2 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 2
General physical health deterioration (General disorders) | 0 | 0 | 11 | 2
Implant site haemorrhage (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 2
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 2 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 2
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis orbital (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 2 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 6 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Adrenal gland injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Eastern Cooperative Oncology Group perfomance worsened (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 3 | 2
Liver function test abnormal (Investigations) | 1 | 0 | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Radiculitis (Nervous system disorders) | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0
Spinal cord paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 4 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 2 | 0
Renal injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Haemorrhagic ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Device dislocation (General disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0
Urethral meatus stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tivantinib 240 mg BID Cohort (N=28) | Placebo Matching 240 mg BID Cohort (N=15) | Tivantinib 120 mg BID Cohort (N=225) | Placebo Matching 120 mg BID Cohort (N=114)
Anaemia (Blood and lymphatic system disorders) | 11 | 2 | 42 | 17
Neutropenia (Blood and lymphatic system disorders) | 15 | 2 | 28 | 5
Bradycardia (Cardiac disorders) | 3 | 0 | 31 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 12 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 11 | 8
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 47 | 32
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 26 | 15
Ascites (Gastrointestinal disorders) | 6 | 7 | 46 | 24
Constipation (Gastrointestinal disorders) | 1 | 1 | 29 | 14
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 50 | 17
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 12 | 8
Nausea (Gastrointestinal disorders) | 4 | 1 | 50 | 13
Vomiting (Gastrointestinal disorders) | 2 | 0 | 26 | 13
Asthenia (General disorders) | 8 | 2 | 48 | 25
Fatigue (General disorders) | 1 | 4 | 58 | 31
General physical health deterioration (General disorders) | 0 | 1 | 15 | 5
Oedema peripheral (General disorders) | 7 | 1 | 54 | 19
Pyrexia (General disorders) | 6 | 1 | 28 | 15
Nasopharyngitis (Infections and infestations) | 0 | 0 | 9 | 7
Alanine aminotransferase increased (Investigations) | 1 | 2 | 8 | 7
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 14 | 10
Blood bilirubin increased (Investigations) | 1 | 0 | 12 | 6
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 36 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 19 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 19 | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 8 | 8
Dizziness (Nervous system disorders) | 1 | 1 | 16 | 3
Headache (Nervous system disorders) | 0 | 0 | 13 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 32 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 22 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 24 | 21
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 9 | 6
Hypertension (Vascular disorders) | 0 | 1 | 19 | 5
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 5 | 5
Myocardial infarction (Cardiac disorders) | 2 | 0 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 4 | 3
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Haematemesis (Gastrointestinal disorders) | 2 | 0 | 1 | 2
Haemorrhage ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 3 | 2
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 2 | 6 | 4
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 0 | 7 | 3
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Device dislocation (General disorders) | 0 | 1 | 0 | 0
Disease progression (General disorders) | 2 | 0 | 1 | 0
Oedema (General disorders) | 1 | 1 | 1 | 4
Pain (General disorders) | 1 | 1 | 4 | 2
Hepatic failure (Hepatobiliary disorders) | 1 | 2 | 5 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 6 | 3
Jaundice (Hepatobiliary disorders) | 0 | 2 | 6 | 4
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 3
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 8 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 6 | 5
Blood creatinine increased (Investigations) | 0 | 2 | 3 | 3
Blood uric acid increased (Investigations) | 1 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 5 | 3
Lymphocyte count decreased (Investigations) | 0 | 1 | 3 | 0
Platelet count decreased (Investigations) | 5 | 1 | 5 | 5
Weight decreased (Investigations) | 0 | 1 | 11 | 3
Weight increased (Investigations) | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 7 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 6 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 8 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 11 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 5 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 9 | 5
Encephalopathy (Nervous system disorders) | 0 | 1 | 3 | 3
Paraesthesia (Nervous system disorders) | 0 | 1 | 3 | 1
Bradyphrenia (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 10 | 5
Urethral meatus stenosis (Psychiatric disorders) | 0 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 0 | 5 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Bleeding varicose vein (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 3 | 5
Intra-abdominal haematoma (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT01755767/Prot_SAP_000.pdf